CLINICAL TRIAL: NCT06339658
Title: ICG vs Blue Patent as a Tracer in the Performance of TAD in Patients With cN1 Breast Carcinoma After Neoadjuvant Chemotherapy
Brief Title: ICG vs Blue Patent for TAD in cN1 Breast Carcinoma After Neoadjuvant Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Amparo Garcia-Tejedor, Principal Investigator, Hospital Universitari de Bellvitge
Other Study IDs: TAD-ICG
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Axillary Metastases
MeSH Terms: conditions — Breast Neoplasms | interventions — DAT protocol 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Indocianine Green (ICG): ICG tracer
  Interventions: Procedure: Targeted axillary dissection (TAD) by ICG
- Blue patent: Blue patent tracer
  Interventions: Procedure: Targeted axillary dissection (TAD) by Blue patent

INTERVENTIONS:
Procedure: Targeted axillary dissection (TAD) by ICG — Use of ICG during the targeted axillary dissection (TAD)
  Groups: Indocianine Green (ICG)
Procedure: Targeted axillary dissection (TAD) by Blue patent — Use of Blue patent during the targeted axillary dissection (TAD)
  Groups: Blue patent

SUMMARY:
To validate the use of ICG as a tracer during TAD in patients with cN1 breast carcinoma after neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
This patient registry is designed to prospectively collect standardized clinical, imaging, surgical, and pathological data from patients with cN1 breast carcinoma undergoing targeted axillary dissection (TAD) following neoadjuvant chemotherapy, using indocyanine green (ICG) as a lymphatic tracer.

To ensure data quality and consistency the following procedures and quality control measures will be implemented:

Standardized Case Report Forms (CRFs):

All data will be recorded using electronic CRFs developed specifically for the registry. These forms are structured to capture relevant demographic, clinical, radiological, surgical, and pathological variables, including tracer detection rates, number of retrieved nodes, false-negative rates, and complications.

Center Training and Accreditation:

All participating surgeons and radiologists will receive training on standardized procedures for TAD using ICG, including injection technique, intraoperative fluorescence detection, and specimen handling. Regular inter-institutional meetings will be held to reinforce protocol adherence.

Quality Assurance in Imaging and Pathology:

Lymph node localization procedures (e.g., clip placement, imaging review) and histopathological analyses will follow unified protocols.

Ethics and Patient Confidentiality:

All data will be de-identified and managed in compliance with GDPR and local data protection regulations. Informed consent will be obtained from each participant prior to data inclusion.

Follow-up and Outcome Tracking:

The registry will track short- and mid-term surgical outcomes, including detection rates, surgical complications, and axillary recurrence, ensuring longitudinal quality assessment of the ICG-guided TAD approach.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer cN+ patients who undergo neadjuvant treatment.

Exclusion Criteria:

* Patients in whom there is a contraindication for the use of ICG.
* Patients in whom there is evidence of progression of the disease after neoadjuvant treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer cN+ patients who underwent neadjuvant treatment and will be candidates to perfom a targeted axillay dissection.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate of sentinel lymph node between tracers | 2 years
  Compare the detection rate of sentinel lymph node between ICG and blue patent in cN+ patients after neoadjuvant treatment

SECONDARY OUTCOMES:
Detection rate of SLNB with ICG versus Tc99 | 2 years
  Compare the detection rate of sentinel lymph node between ICG and Tc99 in cN+ patients after neoadjuvant treatment
Adverse effects | 2 years
  Evaluate the adverse effects from the use of each of the tracers

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ortega-Expósito, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided